CLINICAL TRIAL: NCT05870241
Title: Post-Mastectomy Shoulder Pain And Lymphedema Responses To Ga-As Laser Versus Microcurrent Electrical Stimulation
Acronym: PM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Catherine Moanis Labib Botros, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003506
Record Dates: First submitted 2023-05-12; First posted 2023-05-23 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Post Mastectomy Lymphedema
Keywords: post mastectomy; lymphedema; pain; Ga-As Laser; Microcurrent
MeSH Terms: conditions — Breast Cancer Lymphedema; Lymphedema; Pain

STUDY DESIGN:
Intervention Model Description: Ga-As Laser and Microcurrent
Who Masked: Outcomes Assessor
Masking Description: random generator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ga-As Laser (Experimental): the patients will receive Ga-As Laser and traditional therapy three times a week for three months
  Interventions: Other: Ga-As Laser; Other: traditional therapy
- Microcurrent Electrical Stimulation (Experimental): the patients will receive Microcurrent Electrical Stimulation and traditional therapy three times a week for three months
  Interventions: Other: Microcurrent Electrical Stimulation; Other: traditional therapy
- traditional therapy (Active Comparator): the patients will receive traditional therapy three times a week for three months
  Interventions: Other: traditional therapy

INTERVENTIONS:
Other: Ga-As Laser — Patient sits on a chair with back support and the two GA-AS laser ( 5 milli Watts & 904 nm) probe will be applied one on the shoulder tip for 5 minutes and the other application another 5 minutes will be on the center of deltoid muscle. The main power of the laser switch will be turned on. The duration of the treatment will be 10 minutes.
  Arms: Ga-As Laser
Other: Microcurrent Electrical Stimulation — The patient sits on a chair with back support and the two electrodes from Microcurrent 850 unit device will be applied one on the shoulder tip and the other electrode on the center of the deltoid muscle. A wet cloth was placed between the electrode and the patient's skin. An adhesive tape was used to hold the electrode over the treated areas. The main power switch will be turned on. The treatment duration will be for 10 minutes.
  Arms: Microcurrent Electrical Stimulation
Other: traditional therapy — the patients will receive traditional physical therapy in the form of manual lymphatic drainage , compression bandage, exercise to increase lymphatic drainage, skin care. and ROM exercises to improve shoulder mobility

SUMMARY:
the aim of this study is to investigate the effect of GA-AS laser versus microcurrent on post-mastectomy shoulder pain and lymphedema.

DETAILED DESCRIPTION:
Breast cancer is extremely rare before the age of 25. It reaches a high incidence in the decade from 40 to 50 and continuous to increase in the frequency into old age. Mastectomy is the traditional approach to remove the entire breast once the diagnosis was confirmed. The most common cancers are lung cancer in men and breast cancer in women, however despite the large numbers of people affected by cancer there is very little literature on the role of physiotherapists in cancer care. After mastectomy and the accompanying excision or radiation of adjacent axillary lymph nodes a patient is at risk of developing upper extremity lymphedema, shoulder pain and loss of shoulder motion.low-level laser light waves penetrate deeply into the skin, they optimize the immune responses of our blood. This has both anti-inflammatory and immunosuppressive effects. It is a scientific fact that light transmitted to the blood in this way has positive effects throughout the whole body, supplying vital oxygen and energy to every cell .Electrical stimulation is based on the fact that human body has an endogenous bioelectric system that enhances healing of bone fracture, soft tissue lesions and decreasing post-operative pain. The external current may serve to mimic the failed natural bioelectric currents, so that post-operative pain can be inhibited. It was reported that microcurrent electrical neuromuscular stimulation (MENS) is better in enhancing cellular physiology processes than other current of higher amplitude, microcurrent is effective in the management of open wounds, inflammation and pain. sixty patients will be randomly allocated to three groups; first one will receive laser+ traditional therapy, second one will receive microcurrent + traditional therapy and third one will receive traditional therapy three times a week for three months.

ELIGIBILITY:
Inclusion Criteria:

All patients will be female patient. Their ages will be ranged from 40 to 55 years old. All patients will have postmastectomy shoulder pain and lymphedema. All patients will be assessed carefully by the physician before the starting of the study procedures.

All patients will be conscious and ambulant. All patients will have surgical mastectomy on the right breast region (site of the surgical excision is right side).

The common indication of breast mastectomy for all cases will be pathological disorder of the breast (breast cancer).

All patients will receive the same necessary or required drugs and diet regime. All patients in the three groups of the study will receive the same medications (antibiotics and diuretics) (Akai

Exclusion Criteria:

Patients who have other pathological conditions or histories except postmastectomy shoulder pain and lymphedema.

Patients with evidence of local recurrence or distant metastasis will be excluded from the study.

Patient who takes other medications that may affects the results Patients who are not ambulant Patients who have surgical mastectomy on the left side breast region not the right one.

Patients who are not co-operative during assessment and treatment.

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
pain intensity | up to twelve weeks
  pain intensity will be measured by visual analogue scale
Lymphedema volume | up to twelve weeks
  lymphedema volume will be measured by measuring the circumference of each segment of the limb between two consecutive circumferences as a truncated zone. The volume of the segment was calculated as V=h(C12 +C1C2+C22 )/12π, where V is the volume of the segment, C1 and C2 are the circumferences at the ends of the segment, and h is the distance between them (segment length)

CONTACTS AND LOCATIONS:
Locations (1):
- Catherine, Giza, Egypt